CLINICAL TRIAL: NCT00451087
Title: Phase 1 Study: Comparison of Electromechanical Delay Phase 2 Study: Research in Viscoelasticity of Tendon Structures Phase 3 Study: Effects of Exercise Training in the Mechanical Properties
Brief Title: Comparisons of Mechanical Properties of Tendon Structures
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Mei-Hwa Jan / Associate Professor, School and Graduate Institute of Physical Therapy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9561703048
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2006-12

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: mechanical properties; electromechanical delay; viscoelasticity; VMO; patellofemoral pain syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: leg press training
- 2 (Active Comparator)
  Interventions: Procedure: isokinetic training

INTERVENTIONS:
Procedure: leg press training — quadriceps muscle strengthening. 30min/ 3times/ week
  Arms: 1
Procedure: isokinetic training — quadriceps muscle training. 30 min/ 3 times/ week
  Arms: 2

SUMMARY:
We assume the etiology of patellofemoral pain syndrome is related to mechanical properties of tendon structures of the vastus medialis obliquus and vastus lateralis. Consequently, we will measure the electromechanical delay and some viscoelastic parameters of the two muscles. Besides, we will also investigate the effects of exercise training to the mechanical properties of the muscles.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is a common knee disorder. From the literature review, one may find inconsistent results among different research or clinical studies on the effect of therapeutic exercise for the patients with PFPS. A possible reason for the disagreement might be lack of a clear etiology of patellofemoral pain. At present, the most widely accepted concept for the genesis of patellofemoral pain is abnormal lateral tracking of the patella. One factor that causes this maltracking is soft tissue imbalance around the patella. Previous studies demonstrating the inconsistency of the amplitude of muscle activity and the timing of muscle firing for vastus medialis obliquus (VMO) and vastus lateralis (VL) may contribute to the imbalance of soft tissue. Another neuromuscular condition, however, the electromechanical delay of VMO and VL in patents with PFPS was not investigated extensively. We hypothesized that people with PFPS would have longer electromechanical delay of VMO than that of VL. The objective of this three-year project is to compare the electromechanical delay of VMO with that of VL in people with PFPS for the first year. In the second year, we will further investigate the viscoelastic properties of tendon structures, the key components induced this electromechanical delay, of VMO and VL in vivo. In the last year, we will research the effect of an exercise program on the mechanical properties of VMO and VL in people with PFPS.We expect to recruit 30 patients with PFPS as an experimental group and 30 healthy individuals as a control group in the both first and second years. In the third year, we will recruit 60 patients with PFPS, 30 of them to receive a specific exercise program and the others are in the control group.

The evoked electromechanical delay of VMO is defined as the time interval between the time when VMO receiving an electrical stimulation and the onset time of patellar movement due to the VMO contraction. The viscoelastic properties of tendon structures are investigated by an ultrasonographic study under voluntary contraction conditions. The torque output during isometric knee extension at 80° of flexion is measured by a dynamometer. The subject is instructed to produce a gradually increasing force from relaxed status to maximal voluntary contraction within 5 seconds, followed by a gradual relaxation also within 5 seconds. Simultaneously, the elongation of the deep aponeurosis of the VMO or VL is caught by the ultrasonic image which is synchronized with the torque signal by a clock timer for subsequent analysis. The stiffness, Young's modulus and hysteresis of the tendon structures are calculated to represent its viscoelastic properties.

Finally, the subject is prescribed an 8-week exercise program by EN-dynamic machine to perform knee extension from 45° to 0° of flexion. The training outcome is assessed with electromechanical delay of VMO and VL. And we will also investigate the effect of the exercise program on the mechanical properties of tendon structures.

ELIGIBILITY:
Inclusion Criteria:

1. Below 50 years old.
2. Subjects have at least two of five conditions of knee pain: to squat down, to go or down stairs, to keep prolong sitting position, to be palpated the joint cartilage of patella, to be test by Clark sign.
3. Subjects have the symptoms for 3 months at least.

Exclusion Criteria:

1. Subjects have the other knee disorder in addition to PFPS.
2. Subjects had ever received operations of knee in past 3 months.
3. Subjects have neurological disease.

Max Age: 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-03 (Actual); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
electromechanical delay | minisecond

SECONDARY OUTCOMES:
quadriceps muscle force | second
the displacement of deep aponeurosis of vasti muscles | second

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hwa Jan, Master, Study Director — School and Graduate Institude of Physical Therapy,NTU
Locations (1):
- Kinesiology Laboratory, Taipei, Taiwan

REFERENCES:
- [Background] Cowan SM, Hodges PW, Bennell KL, Crossley KM. Altered vastii recruitment when people with patellofemoral pain syndrome complete a postural task. Arch Phys Med Rehabil. 2002 Jul;83(7):989-95. doi: 10.1053/apmr.2002.33234. PMID 12098160
- [Result] Kubo K, Kanehisa H, Kawakami Y, Fukunaga T. Elastic properties of muscle-tendon complex in long-distance runners. Eur J Appl Physiol. 2000 Feb;81(3):181-7. doi: 10.1007/s004210050028. PMID 10638375
- [Derived] Chen HY, Chien CC, Wu SK, Liau JJ, Jan MH. Electromechanical delay of the vastus medialis obliquus and vastus lateralis in individuals with patellofemoral pain syndrome. J Orthop Sports Phys Ther. 2012 Sep;42(9):791-6. doi: 10.2519/jospt.2012.3973. Epub 2012 Aug 2. PMID 22951377